CLINICAL TRIAL: NCT04788238
Title: Dual-Task Zumba Gold for Improving the Cognition of Community-Dwelling Older Adults With Mild Cognitive Impairment: A Pilot Randomized Controlled Trial
Brief Title: Dual-Task Zumba Gold for Improving the Cognition of Older Adults With MCI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, Dr Angela Leung, Associate Professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: HSEARS20200717002
Record Dates: First submitted 2021-02-25; First posted 2021-03-09 (Actual); Last update posted 2022-02-04 (Actual); Status verified 2022-01

CONDITIONS: Mild Cognitive Impairment
Keywords: dual-task; Zumba Gold; mild cognitive impairment; dementia risk reduction
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: Participants will be equally allocated to the intervention and control group, following a randomization schedule generated by an independent statistician who has no access to the subjects. The randomization list will be sealed in sequentially numbered opaque envelopes. Participants will be informed of the group allocation after the submission of written consent and completion of the baseline assessments.
Who Masked: Outcomes Assessor
Masking Description: Outcome assessors and data analysts will be blinded to the group allocation until the whole data analyses are completed. They will also not be involved in any part of the treatment administration. Furthermore, participants will be advised not to disclose their group assignment during data collection.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Participants in the intervention arm will participate in the dual-task Zumba Gold (DTZ) program. They will be grouped into 10 participants per class.
  Interventions: Behavioral: Dual-Task Zumba Gold
- Control group (No Intervention): Participants in the control group will receive health education about dementia risk reduction provided by community health nurses.

INTERVENTIONS:
Behavioral: Dual-Task Zumba Gold — Dual-Task Zumba Gold is a 12-week program to be conducted thrice weekly for 45-60 minutes. The intervention involves the concurrent performance of cognitive tasks and physical movements during specific parts of the dance. The activity will begin with warm-up and end with cool-down periods, at 5 to 10 minutes each. Orientation training will be done during the warm-up period, by asking questions to participants about time, place, and person. In the actual dance (30 to 40 minutes), the following domains will be trained: executive function (forward and backward serial counting); perceptual-motor ability (performing arm clock positions based on instructions); memory (forward and backward repetition of number/word series), and attention (forward and backward spelling of 3- to 5-letter words). The cool-down period will incorporate memory training by reminding the participants to summarize the activities performed.
  Arms: Intervention group

SUMMARY:
The study aims to assess the preliminary efficacy of a Dual-Task Zumba Gold (DTZ) intervention that will support physical and cognitive training among community-dwelling persons with mild cognitive impairment (MCI). A 12-week Dual-Task Zumba Gold (DTZ) intervention will be implemented among 30 participants with MCI in the treatment group, while health education will be provided to another 30 subjects allocated in the control group. Changes in global cognitive function, together with the quality of life, mood, functional mobility, and bodily measures, will be re-assessed after the 12-week intervention and a 6-week follow-up period. Quantitative and qualitative methods will also be employed to assess the feasibility and acceptability outcomes of the study.

DETAILED DESCRIPTION:
Background: Dementia risk reduction is considered a public health priority. However, there is a paucity of related interventions among low- and middle-income countries (LMICs), such as the Philippines, despite the higher number of dementia cases in these regions. Meanwhile, individuals with mild cognitive impairment (MCI), being at risk for dementia, are important targets for interventions to promote cognitive health.

The enrichment of physical activities with cognitive exercises, known as dual-task training, is an innovative approach that has been noted to potentially improve cognitive outcomes in persons with MCI. Zumba is a popular dance worldwide, which combines rhythmic aerobic steps and whole-body movements. It has a modified version for older adults, called Zumba Gold, but information about its effects on older people is limited.

Literature states that ensuring sufficient cognitive load in complex motor activities is important to achieve significant and superior cognitive outcomes. Dual-Task Zumba Gold (DTZ), an intervention combining Zumba Gold and simultaneous cognitive training, and is a novel and inexpensive non-pharmacological intervention that may enhance the cognition of persons at risk for dementia. However, its feasibility and potential efficacy among older people with MCI are unknown.

Objectives of the Study: There are two objectives in this study: (1) To determine the feasibility and acceptability of a Dual-Task Zumba Gold (DTZ) intervention among community-dwelling individuals with MCI. (2) To investigate the preliminary efficacy of the DTZ intervention in improving the cognitive function among the recruited participants with MCI.

Methods: This is a mixed-method pilot study, involving quantitative and qualitative methods to evaluate the study outcomes. The proposed 12-week DTZ intervention will be conducted three times/week for 45-60 minutes among individuals with MCI. Cognitive domains of executive function, visuospatial ability, memory, and complex attention will be stimulated through mental exercises which will be performed concurrently with the dance steps during particular sequences of the Zumba Gold dance.

Sixty participants will be recruited, and then randomly allocated to treatment (DTZ) and control groups (health education). The feasibility of the intervention will be assessed by participant recruitment and retention rate, adherence rate, and implementation fidelity. Acceptability will be evaluated quantitatively via self-report attitudes towards the intervention. Moreover, qualitative data will be collected via focus group discussions to obtain their feedback toward the intervention.

Changes in cognitive function will be assessed as the primary outcomes, to be measured via the following tools: Montreal Cognitive Assessment (MoCA-P) for global cognition; Trail Making Tests A and B (TMT A & B) for executive functioning; Digit Span Test (DST) and MoCA-Memory Index Score (MoCA-MIS) for memory. Secondary outcomes to be evaluated include quality of life (Perceived Well-being Scale), mood (Geriatric Depression Scale-Short Form), functional mobility (Short Physical Performance Battery), and bodily measures (blood pressure, body mass index, and waist circumference).

Content analysis will be utilized to analyze qualitative data from the interviews. Meanwhile, descriptive statistics, Chi-square test, and independent t-test will be used to analyze the subjects' characteristics and compare the two groups at baseline. Generalized estimating equations (GEE) will be used to determine the intervention's preliminary efficacy at the post-treatment period.

ELIGIBILITY:
Inclusion Criteria:

* subjective report/concern about changes in memory or cognition
* objective cognitive impairment, based on Montreal Cognitive Assessment (MoCA) score of ≤25
* absence of diagnosis of dementia or Alzheimer's disease
* normal function in daily activities, via Katz ADL scale score of 6
* ambulatory, without the need to use assistive devices
* able to read/communicate in the Filipino/English language

Exclusion Criteria:

* medical diagnosis of any form of neurological or psychiatric disorder
* uncontrolled or severe heart condition, cancer, major musculoskeletal disorder, psychiatric condition, serious hearing/visual impairment, or any condition that would limit study safety; or being at risk for adverse events to PA participation, assessed via the revised Physical Activity Readiness Questionnaire (rPARQ)
* intake of medications such as anti-depressants, sedatives, or anti-epileptics that may affect cognition
* participation in any organized physical activity program in the past 3 months

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-03-29 (Actual); Primary Completion 2021-10-15 (Actual); Study Completion 2022-08-31 (Estimated)

PRIMARY OUTCOMES:
Changes in Montreal Cognitive Assessment score (from baseline to 18 weeks follow-up) | Baseline; 12 weeks; 18 weeks
  Montreal Cognitive Assessment (MoCA) evaluates global cognition by involving multiple domains such as attention, memory, language, visuospatial skills, abstraction, calculation, and orientation. The scores range from 0 to 30, with higher scores indicating better cognitive performance.
Changes in Trail Making Test Part A (from baseline to 18 weeks follow-up) | Baseline; 12 weeks; 18 weeks
  Trail Making Test Part A is a time-based examination that requires individuals to connect randomly arranged numbers following the correct sequence. The time limit for this test is up to 150 seconds, and shorter duration pertains to better processing speed.
Changes in Trail Making Test Part B (from baseline to 18 weeks follow-up) | Baseline; 12 weeks; 18 weeks
  Trail Making Test Part B is a time-based examination that requires individuals to connect randomly arranged numbers and letters following the correct and alternating sequence. The time limit for this test is up to 300 seconds, and shorter duration pertains to better executive function.
Changes in Digit Span test (from baseline to 18 weeks follow-up) | Baseline; 12 weeks; 18 weeks
  In Digit Span Test, numbers are read to the participant at a rate of one per second and then later asked to repeat them in a forward and backward manner. Scores range from 0 - 14 and higher scores indicate better short-term memory.
Changes in the MoCA-Memory Index score (from baseline to 18 weeks follow-up) | Baseline; 12 weeks; 18 weeks
  The Memory Index Score of the Montreal Cognitive Assessment (MoCA-MIS) ranges from 0-15, which is based on free delayed recall, category cued recall, and multiple choice cued recall. Higher scores indicate better delayed recall ability.

SECONDARY OUTCOMES:
Changes in quality of life using Perceived Well-Being Scale (from baseline to 18 weeks follow-up) | Baseline; 12 weeks; 18 weeks
  The Perceived Well-Being Scale (PWB) assesses older adults' quality of life in the physical and psychological domains, using a 14-item tool with a 7-point Likert scale. Its scores range from 14-98, and higher values pertain to higher quality of life.
Changes in mood using Geriatric Depression Scale-Short Form (from baseline to 18 weeks follow-up) | Baseline; 12 weeks; 18 weeks
  The Geriatric Depression Scale-Short Form (GDS-SF) is a 15-item instrument which is answered dichotomously by 'yes' or 'no' responses. Scores range from 0-15, with lower scores pertaining to better emotional status.
Changes in functional mobility using Short Physical Performance Battery (from baseline to 18 weeks follow-up) | Baseline; 12 weeks; 18 weeks
  The Short Physical Performance Battery (SPPB) measures timed performance on three tasks (standing balance, gait speed, and rising from a chair) to derive a score from 0-12. Higher scores indicate better functional mobility.
Changes in blood pressure (from baseline to 18 weeks follow-up) | Baseline; 12 weeks; 18 weeks
  Blood pressure will reflect systolic and diastolic measures, and will be assessed through calibrated blood pressure monitors.
Changes in body-mass index (from baseline to 18 weeks follow-up) | Baseline; 12 weeks; 18 weeks
  Body mass index will be reported in kg/m^2, by obtaining the participants' weight (in kilograms) and height (in meters) via a Detecto scale.
Changes in waist circumference (from baseline to 18 weeks follow-up) | Baseline; 12 weeks; 18 weeks
  Waist circumference will be measured in centimeters via tape measure.

CONTACTS AND LOCATIONS:
Overall Officials: Angela Leung, PhD, Principal Investigator — The Hong Kong Polytechnic University
Locations (1):
- Municipality of Plaridel, Plaridel, Bulacan, Philippines

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abbott JH. The distinction between randomized clinical trials (RCTs) and preliminary feasibility and pilot studies: what they are and are not. J Orthop Sports Phys Ther. 2014 Aug;44(8):555-8. doi: 10.2519/jospt.2014.0110. No abstract available. PMID 25082389
- [Background] American College of Sports Medicine; Chodzko-Zajko WJ, Proctor DN, Fiatarone Singh MA, Minson CT, Nigg CR, Salem GJ, Skinner JS. American College of Sports Medicine position stand. Exercise and physical activity for older adults. Med Sci Sports Exerc. 2009 Jul;41(7):1510-30. doi: 10.1249/MSS.0b013e3181a0c95c. PMID 19516148
- [Background] Barcelos N, Shah N, Cohen K, Hogan MJ, Mulkerrin E, Arciero PJ, Cohen BD, Kramer AF, Anderson-Hanley C. Aerobic and Cognitive Exercise (ACE) Pilot Study for Older Adults: Executive Function Improves with Cognitive Challenge While Exergaming. J Int Neuropsychol Soc. 2015 Nov;21(10):768-79. doi: 10.1017/S1355617715001083. PMID 26581789
- [Background] Cardinal BJ, Esters J, Cardinal MK. Evaluation of the revised physical activity readiness questionnaire in older adults. Med Sci Sports Exerc. 1996 Apr;28(4):468-72. doi: 10.1097/00005768-199604000-00011. PMID 8778552
- [Background] Dalleck LC, Roos KA, Byrd BR, Weatherwax RM. Zumba Gold((R)): Are The Physiological Responses Sufficient to Improve Fitness in Middle-Age to Older Adults? J Sports Sci Med. 2015 Aug 11;14(3):689-90. eCollection 2015 Sep. No abstract available. PMID 26336358
- [Background] Diamond A, Ling DS. Conclusions about interventions, programs, and approaches for improving executive functions that appear justified and those that, despite much hype, do not. Dev Cogn Neurosci. 2016 Apr;18:34-48. doi: 10.1016/j.dcn.2015.11.005. Epub 2015 Dec 7. PMID 26749076
- [Background] Dominguez JC, Orquiza MG, Soriano JR, Magpantay CD, Esteban RC, Corrales ML, Ampil ER. Adaptation of the Montreal Cognitive Assessment for elderly Filipino patients. East Asian Arch Psychiatry. 2013 Sep;23(3):80-5. PMID 24088400
- [Background] Gheysen F, Poppe L, DeSmet A, Swinnen S, Cardon G, De Bourdeaudhuij I, Chastin S, Fias W. Physical activity to improve cognition in older adults: can physical activity programs enriched with cognitive challenges enhance the effects? A systematic review and meta-analysis. Int J Behav Nutr Phys Act. 2018 Jul 4;15(1):63. doi: 10.1186/s12966-018-0697-x. PMID 29973193
- [Background] Guralnik JM, Simonsick EM, Ferrucci L, Glynn RJ, Berkman LF, Blazer DG, Scherr PA, Wallace RB. A short physical performance battery assessing lower extremity function: association with self-reported disability and prediction of mortality and nursing home admission. J Gerontol. 1994 Mar;49(2):M85-94. doi: 10.1093/geronj/49.2.m85. PMID 8126356
- [Background] Katz S. Assessing self-maintenance: activities of daily living, mobility, and instrumental activities of daily living. J Am Geriatr Soc. 1983 Dec;31(12):721-7. doi: 10.1111/j.1532-5415.1983.tb03391.x. PMID 6418786
- [Background] Kayama H, Okamoto K, Nishiguchi S, Yamada M, Kuroda T, Aoyama T. Effect of a Kinect-based exercise game on improving executive cognitive performance in community-dwelling elderly: case control study. J Med Internet Res. 2014 Feb 24;16(2):e61. doi: 10.2196/jmir.3108. PMID 24565806
- [Background] Lauenroth A, Ioannidis AE, Teichmann B. Influence of combined physical and cognitive training on cognition: a systematic review. BMC Geriatr. 2016 Jul 18;16:141. doi: 10.1186/s12877-016-0315-1. PMID 27431673
- [Background] Luettgen M, Foster C, Doberstein S, Mikat R, Porcari J. Zumba((R)): is the "fitness-party" a good workout? J Sports Sci Med. 2012 Jun 1;11(2):357-8. eCollection 2012. No abstract available. PMID 24137072
- [Background] McIsaac TL, Lamberg EM, Muratori LM. Building a framework for a dual task taxonomy. Biomed Res Int. 2015;2015:591475. doi: 10.1155/2015/591475. Epub 2015 Apr 19. PMID 25961027
- [Background] Moreau D, Morrison AB, Conway AR. An ecological approach to cognitive enhancement: complex motor training. Acta Psychol (Amst). 2015 May;157:44-55. doi: 10.1016/j.actpsy.2015.02.007. Epub 2015 Feb 25. PMID 25725192
- [Background] Nasreddine ZS, Phillips NA, Bedirian V, Charbonneau S, Whitehead V, Collin I, Cummings JL, Chertkow H. The Montreal Cognitive Assessment, MoCA: a brief screening tool for mild cognitive impairment. J Am Geriatr Soc. 2005 Apr;53(4):695-9. doi: 10.1111/j.1532-5415.2005.53221.x. PMID 15817019
- [Background] Petersen RC, Caracciolo B, Brayne C, Gauthier S, Jelic V, Fratiglioni L. Mild cognitive impairment: a concept in evolution. J Intern Med. 2014 Mar;275(3):214-28. doi: 10.1111/joim.12190. PMID 24605806
- [Background] Reker GT, Wong PTP. Psychological and Physical Well-Being in the Elderly: The Perceived Well-Being Scale (PWB). Can J Aging. 1984;3(1):23-32. doi: 10.1017/S0714980800006437.
- [Background] Sachdev PS, Blacker D, Blazer DG, Ganguli M, Jeste DV, Paulsen JS, Petersen RC. Classifying neurocognitive disorders: the DSM-5 approach. Nat Rev Neurol. 2014 Nov;10(11):634-42. doi: 10.1038/nrneurol.2014.181. Epub 2014 Sep 30. PMID 25266297
- [Background] Sheikh JI, Yesavage JA. Geriatric Depression Scale (GDS): Recent evidence and development of a shorter version. Clin Gerontol. 1986;5(1):165-173. doi: 10.1300/J018v05n01_09.
- [Background] Thompson WR. Worldwide Survey of Fitness Trends for 2013. ACSMs Health Fit J. 2012;16(6):8-17. doi: 10.1249/01.FIT.0000422568.47859.35.
- [Background] Wechsler DA. Manual for the Wechsler Memory Scale-Revised. New York: Psychological Corporation; 1987.
- [Derived] Parial LL, Kor PPK, Sumile EF, Leung AYM. Dual-Task Zumba Gold for Improving the Cognition of People With Mild Cognitive Impairment: A Pilot Randomized Controlled Trial. Gerontologist. 2023 Aug 24;63(7):1248-1261. doi: 10.1093/geront/gnac081. PMID 35679826

DOCUMENTS (1):
  • Informed Consent Form (2021-02-08): https://cdn.clinicaltrials.gov/large-docs/38/NCT04788238/ICF_000.pdf